CLINICAL TRIAL: NCT04064216
Title: Comparison of Cosmesis, Patient Satisfaction and Quality of Life in Patients Undergoing Robot Assisted Versus Conventional Laparoscopic Surgery for Bening Gynecologic Disorders: a Prospective Trial
Brief Title: Comparison of Cosmesis, Patient Satisfaction and Quality of Life in Patients Undergoing Laparoscopic Surgery
Status: Completed | Type: Observational
Sponsor: Acibadem University (Other)
Responsible Party: Principal Investigator, Esra Ozbasli, Ass. Prof., Acibadem University
Other Study IDs: ATADEK-2018/8
Record Dates: First submitted 2019-08-07; First posted 2019-08-21 (Actual); Last update posted 2020-04-13 (Actual); Status verified 2020-04

CONDITIONS: Gynecologic Disease; Cosmesis; Patient Satisfaction; Quality of Life
Keywords: Cosmesis; Laparoscopic surgery; Patient satisfaction; Scar assessment; Quality of life
MeSH Terms: conditions — Genital Diseases, Female; Patient Satisfaction | interventions — Laparoscopy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 9 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Robot assisted laparoscopic surgery: This group will be consisted of patients that will undergo robot assisted laparoscopic surgery for benign gynecologic disorders
  Interventions: Procedure: Laparoscopic surgery
- Conventional laparoscopic surgery: This group will be consisted of patients that will undergo conventional laparoscopic surgery for benign gynecologic disorders
  Interventions: Procedure: Laparoscopic surgery

INTERVENTIONS:
Procedure: Laparoscopic surgery — Patients that will undergo robot assisted laparoscopic surgery and conventional laparoscopic surgery for benign gynecologic disorders will answer 4 questionnaires to assess patient satisfaction, quality of life and cosmesis

SUMMARY:
To compare robot assisted versus conventional laparoscopic surgery performed for bening gynecologic disorders regarding cosmesis, patient satisfaction and quality of life

DETAILED DESCRIPTION:
30 patients undergoing robot assisted laparoscopic surgery for bening gynecologic disorders and 30 patients undergoing conventional laparoscopic surgery for bening gynecologic disorders will be included in the study. All surgeries will be performed in the same hospital by the same surgeon. 6 months after the surgery the patients will be called and will be informed about the trial. After confirming that the questionnaires can be sent to them by e-mail, 4 questionnaires will be sent to the patients via e-mail. To evaluate cosmesis, patient satisfaction and quality of life VAS (visual analogue scale), SF-12 (short form-12) health survey, BIQ (body image questionnaire) and POSAS (the patient and observer scar assessment scale) will be sent to the patients 6 months after the surgery. Patients who have not completed the questionnaires will be called for reminders after 1 week. Patients will be expected to complete the questionnaire completely and accurately.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a diagnosis of being gynecologic disorders
* Patients undergoing conventional laparoscopic surgery
* Patients undergoing robot assisted laparoscopic surgery
* Patients undergoing surgery in our hospital by the same surgeon
* Patients willing to participate in the study

Exclusion Criteria:

* Malignancy
* Requirement of emergency procedure
* Pregnancy
* Visible previous abdominal scars or keloid
* Inability of patient to tolerate Trendelenburg position or pneumoperitoneum
* Patients undergoing surgery by another surgeon or in an another hospital
* Mental impairment that would preclude giving informed consent

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Study Population: 30 patients undergoing robot assisted laparoscopic surgery for bening gynecologic disorders and 30 patients undergoing conventional laparoscopic surgery for bening gynecologic disorders will be included in our study.
Sampling Method: Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2019-07-16 (Actual); Primary Completion 2020-03-16 (Actual); Study Completion 2020-03-16 (Actual)

PRIMARY OUTCOMES:
Patient-perceived cosmesis | 6 months after the surgery
  The primary outcome is to evaluate patient's satisfaction about their laparoscopic incision scars 6 months after the surgery. 6 months after the surgery the patients will be called and will be informed about the trial. After confirming that the questionnaires can be sent to them by e-mail, questionnaires will be sent to the patients. BIQ (body image questionnaire) multiple choice questionnaire to evaluate their scar will be sent to the patients 6 months after the surgery. Patients who have not completed the questionnaires will be called for reminders after 1 week. Patients will be expected to complete the questionnaires completely and accurately.
Patient and observer scar assessment | 6 months after the surgery
  The primary outcome is to evaluate patient's satisfaction about their laparoscopic incision scars 6 months after the surgery. 6 months after the surgery the patients will be called and will be informed about our trial. After confirming that the questionnaires can be sent to them by e-mail, questionnaires will be sent to the patients. POSAS (the patient and observer scar assessment scale) multiple choice questionnaires to evaluate their scar will be sent to the patients 6 months after the surgery. Patients who have not completed the questionnaires will be called for reminders after 1 week. Patients will be expected to complete the questionnaires completely and accurately.

SECONDARY OUTCOMES:
Patient satisfaction | 6 months after the surgery
  To compare patient-reported satisfaction using a scale called visual analogue scale (VAS) will be send to the patients via e-mail. This is a 100-mm long scale with adjectival descriptions at both end positions. There will be a statement explaining what was intended to measure. Participants will be asked to mark the VAS 6 months after the surgery. On this scale 0 representing the worst and 10 the best expected appearance of their scars.
Quality of life after robot assisted versus conventional laparoscopic surgery | 6 months after the surgery
  Quality of life will be measured using SF-12 (short form 12) health questionnaire. This is a 12-Item Short-form Health Survey. 6 months after the surgery the patients will be called and will be informed about our trial. After confirming that the questionnaire can be sent to them by e-mail, questionnaire will be sent to the patients. Patients who have not completed the questionnaires will be called for reminders after 1 week. Patients will be expected to complete the questionnaires completely and accurately.

CONTACTS AND LOCATIONS:
Overall Officials: Mete Gungor, MD,Prof., Study Director — Acıbadem Mehmet Ali Aydınlar University
Locations (1):
- Acibadem Maslak Hospital, Istanbul, Sariyer, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
It will be shared upon request.

REFERENCES:
- [Background] Van Loey NE, Van Son MJ. Psychopathology and psychological problems in patients with burn scars: epidemiology and management. Am J Clin Dermatol. 2003;4(4):245-72. doi: 10.2165/00128071-200304040-00004. PMID 12680803
- [Background] Korolija D, Sauerland S, Wood-Dauphinee S, Abbou CC, Eypasch E, Caballero MG, Lumsden MA, Millat B, Monson JR, Nilsson G, Pointner R, Schwenk W, Shamiyeh A, Szold A, Targarona E, Ure B, Neugebauer E; European Association for Endoscopic Surgery. Evaluation of quality of life after laparoscopic surgery: evidence-based guidelines of the European Association for Endoscopic Surgery. Surg Endosc. 2004 Jun;18(6):879-97. doi: 10.1007/s00464-003-9263-x. Epub 2004 Apr 27. PMID 15108103
- [Background] Corrado G, Calagna G, Cutillo G, Insinga S, Mancini E, Baiocco E, Zampa A, Bufalo A, Perino A, Vizza E. The Patient and Observer Scar Assessment Scale to Evaluate the Cosmetic Outcomes of the Robotic Single-Site Hysterectomy in Endometrial Cancer. Int J Gynecol Cancer. 2018 Jan;28(1):194-199. doi: 10.1097/IGC.0000000000001130. PMID 29040189
- [Background] Yeung PP Jr, Bolden CR, Westreich D, Sobolewski C. Patient preferences of cosmesis for abdominal incisions in gynecologic surgery. J Minim Invasive Gynecol. 2013 Jan-Feb;20(1):79-84. doi: 10.1016/j.jmig.2012.09.008. PMID 23312246